CLINICAL TRIAL: NCT06217965
Title: Evaluation of the Epidemiological and Psychosocial Outcomes of Liver Graft Recipients Transplanted During Childhood
Acronym: EPsyGraft
Status: Recruiting | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/06DEC/498
Record Dates: First submitted 2023-11-20; First posted 2024-01-23 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — The study will involve patients completing a questionnaire on a secure online platform (such as RedCap)

SUMMARY:
The main objective of this study is to better characterize the adult population with a history of liver transplantation in pediatric age. In this context, the investigators will use a questionnaire to assess the participants social environment and lifestyle habits and validated scales to assess their alcohol consumption and anxiety levels.

Secondly, the investigators would like to assess the participants knowledge of their disease, their experience of the transition period from pediatrics to adult medicine, and their compliance with medication.

DETAILED DESCRIPTION:
Outcomes after pediatric liver transplantation have improved in recent years, thanks to improvements in surgical techniques, immunosuppressive drugs and postoperative management in pediatric hepatology departments. For some diseases, transplantation has become the only way to save the lives of these children, or to ensure them a better quality of life.

Indications for pediatric liver transplantation can be categorized as follows: Cholestatic condition, hepatitis, metabolic diseases, tumors and orther conditions such as Gestational alloimmune liver disease, drug induced liver diseases, ect.

Short- and long-term complications following liver transplantation have been the subject of numerous studies.

These include mainly biliary and vascular complications, rejection and infections (including EBV viral infections, which can lead to post-transplant lymphoproliferative disorder).

A recent study showed that in the long term, only 32% of children with liver transplants had an "ideal outcome" defined as a first allograft stable on immunosuppression monotherapy, normal growth, and absence of common immunosuppression-induced sequelae.

However, there are few studies on the epidemiological and social outcome of pediatric liver transplantation. Our French colleagues have published in 2008 one of the few studies on the subject, which reports notably that young adults with a history of liver transplants in paediatric age were anxious about their future, had lower alcohol consumption than the general population, but that medication compliance remained a challenge to be improved.

The aim of our research project is to broaden our knowledge of the subject by assessing the epidemiological and social impact of pediatric liver transplantation on French-speaking liver transplant patients followed at the Cliniques Universitaires Saint Luc.

Objective data on these points will enable us to reinforce our prevention and social support measures, and to review our transfer protocols from pediatric to adult medicine.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over 18 years old who received a pediatric liver transplant and who have been followed regularly at the Saint-Luc university clinics is eligible for inclusion in this study provided they speak French/Dutch fluently

Exclusion Criteria:

* patients minor (< 18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients who received liver transplants before the age of 18 (pediatric transplants) and who have been followed regularly at Cliniques universitaires Saint-Luc. These patients must speak French or Dutch.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
assessing the epidemiological and social impact of pediatric liver transplantation | 1 year
  To better characterize the adult population with a history of liver transplantation in pediatric age. In this context, we will use a questionnaire to assess :
  * social environment (level of education, social status, employment, sexual orientation...)
  * lifestyle habits (risk-taking behavior, diet, exercise, weight, height…)
  * validated scales to assess their alcohol consumption and anxiety levels (AUDIT, BDI, STAI)

SECONDARY OUTCOMES:
assessing their knowledge of their disease, their experience of the transition period from pediatrics to adult medicine, and their compliance with medication | 1 year
  to assess by questionnaire their knowledge of :
  * their disease (name, mechanism…)
  * their experience of the transition period from pediatrics to adult medicine (âge, personal experience…)
  * their compliance with medication (number of treatments, gradation of compliance by type of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Stephenne, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Avanie Hippocrate 10, Woluwe-Saint-Lambert, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dommergues JP, Letierce A, Descots C, Debray D. [Medical follow-up, everyday life and actual experience of young adults after liver transplantation in childhood]. Arch Pediatr. 2008 Jun;15(5):855-6. doi: 10.1016/S0929-693X(08)71940-7. No abstract available. French. PMID 18582779
- [Background] Kohli R, Cortes M, Heaton ND, Dhawan A. Liver transplantation in children: state of the art and future perspectives. Arch Dis Child. 2018 Feb;103(2):192-198. doi: 10.1136/archdischild-2015-310023. Epub 2017 Sep 16. PMID 28918383
- [Background] Ng VL, Alonso EM, Bucuvalas JC, Cohen G, Limbers CA, Varni JW, Mazariegos G, Magee J, McDiarmid SV, Anand R; Studies of Pediatric Liver Transplantation (SPLIT) Research Group. Health status of children alive 10 years after pediatric liver transplantation performed in the US and Canada: report of the studies of pediatric liver transplantation experience. J Pediatr. 2012 May;160(5):820-6.e3. doi: 10.1016/j.jpeds.2011.10.038. Epub 2011 Dec 20. PMID 22192813
- [Background] Smith SK, Miloh T. Pediatric Liver Transplantation. Clin Liver Dis. 2022 Aug;26(3):521-535. doi: 10.1016/j.cld.2022.03.010. PMID 35868688